CLINICAL TRIAL: NCT02883452
Title: An Open-label, Randomized, Parallel-Group, Phase I Study to Evaluate Pharmacokinetics, Efficacy and Safety Between Subcutaneous CT-P13 and Intravenous CT-P13 in Patients With Active Crohn's Disease and Active Ulcerative Colitis
Brief Title: A Phase I Study to Evaluate Pharmacokinetics, Efficacy and Safety of CT-P13 Subcutaneous in Patients With Active Crohn's Disease and Ulcerative Colitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT-P13 1.6 (SC); 2016-002124-89 (EudraCT Number)
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Crohn's Disease; Ulcerative Colitis (Part 2 Only)
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative | interventions — CT-P13; Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (6):
- Cohort 1: CT-P13 IV 5 mg/kg (Active Comparator): CT-P13 IV (Infliximab), 5 mg/kg by IV infusion every 8 weeks (Part 1)
  Interventions: Biological: CT-P13
- Cohort 2: CT-P13 SC 120 mg (Experimental): CT-P13 SC (Infliximab), 120 mg by SC injection every 2 weeks (Part 1)
  Interventions: Biological: CT-P13
- Cohort 3: CT-P13 SC 180 mg (Experimental): CT-P13 SC (Infliximab), 180 mg by SC injection every 2 weeks (Part 1)
  Interventions: Biological: CT-P13
- Cohort 4: CT-P13 SC 240 mg (Experimental): CT-P13 SC (Infliximab), 240 mg by SC injection every 2 weeks (Part 1)
  Interventions: Biological: CT-P13
- Arm 1: CT-P13 SC 120/240 mg (Experimental): CT-P13 SC (Infliximab), either 120 mg or 240 mg every 2 weeks by SC injection (Part 2)
  Interventions: Biological: CT-P13
- Arm 2: CT-P13 IV 5 mg/kg (Active Comparator): CT-P13 IV (Infliximab), 5 mg/kg by IV infusion every 8 weeks up to Week 22. CT-P13 IV was switched to either 120 mg or 240 mg of CT-P13 SC (Infliximab) treatment, and further doses with CT-P13 SC were given up to Week 54. (Part 2)
  Interventions: Biological: CT-P13

INTERVENTIONS:
Biological: CT-P13 — CT-P13 (5 mg/kg) by IV infusion administered as a 2-hour IV infusion per dose every 8 weeks (Part 1)
  Other Names: Infliximab
  Arms: Cohort 1: CT-P13 IV 5 mg/kg
Biological: CT-P13 — CT-P13 (120 mg) by single SC injection every 2 weeks (Part 1)
  Other Names: Infliximab
  Arms: Cohort 2: CT-P13 SC 120 mg
Biological: CT-P13 — CT-P13 (180 mg) by double SC 90 mg injections every 2 weeks (Part 1)
  Other Names: Infliximab
  Arms: Cohort 3: CT-P13 SC 180 mg
Biological: CT-P13 — CT-P13 (240 mg) by double SC 120 mg injections every 2 weeks (Part 1)
  Other Names: Infliximab
  Arms: Cohort 4: CT-P13 SC 240 mg
Biological: CT-P13 — CT-P13 (120 mg) by single SC injection every 2 weeks in patients with body weight less than 80 kg, and CT-P13 (240 mg) by double SC 120 mg injections in patients with body weight at or above 80 kg based on body weight at Week 6 (Part 2)
  Other Names: Infliximab
  Arms: Arm 1: CT-P13 SC 120/240 mg
Biological: CT-P13 — CT-P13 (5 mg/kg) by IV infusion administered as a 2-hour IV infusion per dose every 8 weeks up to Week 22. From Week 30, CT-P13 (120 mg) by single SC injection every 2 weeks in patients with body weight less than 80 kg, and CT-P13 (240 mg) by double SC 120 mg injections in patients with body weight at or above 80 kg based on body weight at Week 30 (Part 2)
  Other Names: Infliximab
  Arms: Arm 2: CT-P13 IV 5 mg/kg

SUMMARY:
Phase 1 randomized, open-label, multicenter, parallel-group study designed to evaluate efficacy, pharmacokinetics and safety between CT-P13 subcutaneous (SC) and CT-P13 intravenous (IV) in patients with active Crohn's Disease (CD) and active Ulcerative Colitis (UC).

DETAILED DESCRIPTION:
A new subcutaneous infliximab formulation is developed by Celltrion, Inc. as an alternative to the intravenous regimen where subcutaneous infliximab injection typically takes less than 2 minutes. The availability of a subcutaneous formulation of infliximab would increase the treatment options available to patients, particularly those wishing to self-administer their therapy. This Phase 1 randomized, open-label, multicenter, parallel-group study is designed to evaluate efficacy, pharmacokinetics and safety between CT-P13 SC and CT-P13 IV in patients with active CD and active UC.

ELIGIBILITY:
Inclusion Criteria:

* Patient has active Crohn's disease with a score on the Crohn's disease activity index between 220 and 450 points.
* Patient has active Ulcerative colitis as defined by a total Mayo score between 6 and 12 points (Part 2 only).

Exclusion Criteria:

* Patient who has previously received a biological agent for the treatment of CD and UC and/or a tumor necrosis factor-alpha (TNFα) inhibitor for the treatment of other disease
* Patient who has allergies to any of the excipients of infliximab or any other murine and/or human proteins or patient with a hypersensitivity to immunoglobulin product
* Patient who has a current or past history of infection with HIV, hepatitis B, or hepatitis C (carriers of hepatitis B and hepatitis C are not permitted to enrol into the study, but past hepatitis B resolved can be enrolled)
* Patient who has acute infection requiring oral antibiotics within 2 weeks or parenteral injection of antibiotics within 4 weeks prior to the first administration of the study drug, other serious infection within 6 months prior to the first administration of study drug or recurrent herpes zoster or other chronic or recurrent infection within 6 weeks prior to the first administration of the study drug
* Patient who has an indeterminate result for interferon-γ release assay (IGRA) or latent tuberculosis (TB) at Screening. For Part 2, if IGRA result is indeterminate at Screening, 1 retest will be possible during the screening. If the repeated IGRA result is negative, the patient can be included in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MoonSun Choi, Study Director — Celltrion
Locations (1):
- Yeungnam University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] D'Haens G, Reinisch W, Schreiber S, Cummings F, Irving PM, Ye BD, Kim DH, Yoon S, Ben-Horin S. Subcutaneous Infliximab Monotherapy Versus Combination Therapy with Immunosuppressants in Inflammatory Bowel Disease: A Post Hoc Analysis of a Randomised Clinical Trial. Clin Drug Investig. 2023 Apr;43(4):277-288. doi: 10.1007/s40261-023-01252-z. Epub 2023 Apr 1. PMID 37004656
- [Derived] Schreiber S, Ben-Horin S, Leszczyszyn J, Dudkowiak R, Lahat A, Gawdis-Wojnarska B, Pukitis A, Horynski M, Farkas K, Kierkus J, Kowalski M, Lee SJ, Kim SH, Suh JH, Kim MR, Lee SG, Ye BD, Reinisch W. Randomized Controlled Trial: Subcutaneous vs Intravenous Infliximab CT-P13 Maintenance in Inflammatory Bowel Disease. Gastroenterology. 2021 Jun;160(7):2340-2353. doi: 10.1053/j.gastro.2021.02.068. Epub 2021 Mar 5. PMID 33676969

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For Part 1, participants were screened from 21 study centers in 9 countries and were enrolled from 20 study centers in 9 countries. For Part 2, participants were screened from 62 study centers in 16 countries and were enrolled from 50 study centers in 15 countries.
Pre-assignment Details: For Part 1, a total of 55 CD patients were screened, 45 patients were enrolled (10 screening failures) and 44 patients were randomized. For Part 2, a total of 195 CD and UC patients were screened, 136 patients were enrolled (59 screening failures) and 131 patients were randomized.
Groups:
- Cohort 1: CT-P13 IV 5 mg/kg (Part 1): Each participant received 2 CT-P13 IV infusions with a 2-week interval at Weeks 0 and 2. Then, this group received further 7 doses of CT-P13 IV 5 mg/kg (Infliximab) by IV infusion at Week 6 and every 8 weeks thereafter up to Week 54.
- Cohort 2: CT-P13 SC 120 mg (Part 1): Each participant received 2 CT-P13 IV infusions with a 2-week interval at Weeks 0 and 2. Then, this group received CT-P13 SC 120 mg (Infliximab) with a 2-week interval from Week 6. The dose of SC 120 mg was adjusted to SC 120 or 240 mg every 2 weeks based on their body weight after Week 30 in applicable patients in Cohort 2: CT-P13 SC 120 mg.
- Cohort 3: CT-P13 SC 180 mg (Part 1): Each participant received 2 CT-P13 IV infusions with a 2-week interval at Weeks 0 and 2. Then, this group received CT-P13 SC 180 mg (Infliximab) with a 2-week interval from Week 6. The dose of SC 180 mg was adjusted to SC 120 or 240 mg every 2 weeks based on their body weight after Week 30 in applicable patients in Cohort 3: CT-P13 SC 180 mg.
- Cohort 4: CT-P13 SC 240 mg (Part 1): Each participant received 2 CT-P13 IV infusions with a 2-week interval at Weeks 0 and 2. Then, this group received CT-P13 SC 240 mg (Infliximab) with a 2-week interval from Week 6. The dose of SC 240 mg was adjusted to SC 120 or 240 mg every 2 weeks based on their body weight after Week 30 in applicable patients in Cohort 4: CT-P13 SC 240 mg.
- Arm 1: CT-P13 SC 120/240 mg (Part 2): Each participant received 2 CT-P13 IV infusions with a 2-week interval at Weeks 0 and 2. Then, this group received CT-P13 SC (Infliximab) either 120 mg or 240 mg from Week 6 to Week 54 based on their body weight at Week 6 (CT-P13 SC 120 mg for patients < 80 kg; CT-P13 SC 240 mg for patients ≥ 80 kg).
- Arm 2: CT-P13 IV 5 mg/kg (Part 2): Each participant received 2 CT-P13 IV infusions with a 2-week interval at Weeks 0 and 2. Then, this group received CT-P13 IV 5 mg/kg (Infliximab) by IV infusion with a 8-week interval from Week 6 up to Week 22 (Weeks 6, 14 and 22). CT-P13 IV was switched to either 120 mg or 240 mg of CT-P13 SC treatment based on their body weight at Week 30 (CT-P13 SC 120 mg for patients < 80 kg; CT-P13 SC 240 mg for patients ≥ 80 kg), and further doses with CT-P13 SC were given up to Week 54.
Period: Overall Study
Arm/Group | Cohort 1: CT-P13 IV 5 mg/kg (Part 1) | Cohort 2: CT-P13 SC 120 mg (Part 1) | Cohort 3: CT-P13 SC 180 mg (Part 1) | Cohort 4: CT-P13 SC 240 mg (Part 1) | Arm 1: CT-P13 SC 120/240 mg (Part 2) | Arm 2: CT-P13 IV 5 mg/kg (Part 2)
Started | 13 (This cohort is only for Part 1.) | 11 (This cohort is only for Part 1.) | 12 (This cohort is only for Part 1.) | 8 (This cohort is only for Part 1.) | 66 (This arm is for Part 2. All of the patients in Part 2 were screened only for Part 2.) | 65 (This arm is for Part 2. All of the patients in Part 2 were screened only for Part 2.)
Completed | 8 | 9 | 7 | 6 | 55 | 50
Not Completed | 5 | 2 | 5 | 2 | 11 | 15
Not completed — Withdrawal by Subject | 1 | 1 | 3 | 0 | 2 | 5
Not completed — Disease progression | 1 | 0 | 0 | 1 | 4 | 5
Not completed — Adverse Event | 2 | 1 | 1 | 1 | 1 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 4 | 1
Not completed — Death | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All-randomized population: all randomized population consisted of all randomly assigned patients at Week 6, regardless of whether or not any study drug (CT-P13 IV, CT-P13 SC) dosing was completed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: CT-P13 IV 5 mg/kg (Part 1) | Cohort 2: CT-P13 SC 120 mg (Part 1) | Cohort 3: CT-P13 SC 180 mg (Part 1) | Cohort 4: CT-P13 SC 240 mg (Part 1) | Arm 1: CT-P13 SC 120/240 mg (Part 2) | Arm 2: CT-P13 IV 5 mg/kg (Part 2) | Total
Number analyzed (Participants) | 13 | 11 | 12 | 8 | 66 | 65 | 175
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 3 | 2 | 5
  Between 18 and 65 years | 13 | 10 | 12 | 8 | 59 | 57 | 159
  >=65 years | 0 | 1 | 0 | 0 | 4 | 6 | 11
Age, Continuous [Median (Full Range); unit: years] | 34.0 [21 to 62] | 33.0 [22 to 67] | 38.5 [22 to 60] | 42.0 [22 to 53] | 33.0 [18 to 69] | 36.0 [18 to 70] | 36.0 [18 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 4 | 4 | 30 | 30 | 80
  Male | 4 | 8 | 8 | 4 | 36 | 35 | 95
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian/Oriental | 2 | 2 | 3 | 2 | 3 | 4 | 16
  White/Caucasian | 11 | 9 | 9 | 6 | 62 | 60 | 157
  Other | 0 | 0 | 0 | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Bosnia and Herzegovina | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Croatia | 3 | 0 | 0 | 1 | 2 | 1 | 3
  Czechia | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Estonia | 0 | 1 | 0 | 0 | 0 | 3 | 3
  Germany | 0 | 0 | 0 | 0 | 4 | 0 | 4
  Hungary | 0 | 0 | 0 | 0 | 5 | 4 | 9
  Israel | 1 | 1 | 2 | 0 | 4 | 6 | 10
  Latvia | 3 | 1 | 2 | 0 | 2 | 6 | 8
  Poland | 0 | 0 | 0 | 0 | 20 | 23 | 43
  Portugal | 0 | 0 | 0 | 0 | 3 | 0 | 3
  Russia | 2 | 3 | 1 | 0 | 15 | 8 | 23
  Slovakia | 1 | 1 | 1 | 1 | 3 | 3 | 6
  South Korea | 2 | 2 | 3 | 2 | 1 | 4 | 5
  Spain | 0 | 0 | 0 | 0 | 3 | 2 | 5
  Ukraine | 1 | 2 | 2 | 4 | 2 | 4 | 6
  Bulgaria | 0 | 0 | 1 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Descriptive Statistics of Area Under the Concentration-time Curve (AUCτ) of Infliximab at Steady State (Part 1)
Description: For Part 1, the primary PK endpoint of the AUCτ at steady state between Week 22 and Week 30 was analyzed in patients who received all doses (full) of study drug up to Week 30 (prior to Week 30) in the PK population. All patients in SC cohorts were randomly assigned at Week 14 in a 1:1 ratio to either of Group A or B for PK monitoring visit period (Week 22 to Week 30). Therefore, AUCτ was calculated at Week 22 for Cohort 1: CT-P13 IV 5 mg/kg, Weeks 22 and 26 for Group A of SC cohorts, and Week 24 and 28 for Group B of SC cohorts.
Time Frame: Week 22, 24, 26 and 28
Population: The PK population consisted of the all-randomized population who received at least one full dose of study drug at Week 6 or thereafter and who had at least one PK concentration result after Week 6 treatment. Among them, patients who received all doses (full) of study drug up to Week 30 (prior to Week 30) were included for primary PK analysis.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Groups:
- Cohort 1: CT-P13 IV 5mg/kg (Part 1): Each participant received 2 CT-P13 IV infusions with a 2-week interval at Weeks 0 and 2. Then, this group received further 7 doses of CT-P13 IV 5 mg/kg (Infliximab) by IV infusion at Week 6 and every 8 weeks thereafter up to Week 54.
Arm/Group | Cohort 1: CT-P13 IV 5mg/kg (Part 1) | Cohort 2: CT-P13 SC 120 mg (Part 1) | Cohort 3: CT-P13 SC 180 mg (Part 1) | Cohort 4: CT-P13 SC 240 mg (Part 1)
Number analyzed (Participants) | 11 | 9 | 11 | 4
hr*ng/mL
  Week 22: number analyzed (Participants) | 11 | 5 | 4 | 1
  Week 22 | 20825679.963 (8432154.3963) | 7821587.111 (3104412.5348) | 12609504.125 (5112454.7748) | 9377712.620
  Week 24: number analyzed (Participants) | 0 | 4 | 6 | 3
  Week 24 |  | 7409271.434 (2062318.5332) | 6736990.881 (6632584.6372) | 14777046.642 (6894029.2838)
  Week 26: number analyzed (Participants) | 0 | 5 | 5 | 1
  Week 26 |  | 8731448.964 (1799009.3658) | 11649915.371 (6140258.9463) | 9721425.240
  Week 28: number analyzed (Participants) | 0 | 4 | 6 | 3
  Week 28 |  | 6589313.495 (984927.8419) | 7038910.791 (6502356.3807) | 14110560.823 (5628122.2174)

2. Primary Outcome: Analysis of Covariance Model (ANCOVA) of Observed Ctrough,week22 (Pre-dose Level at Week 22) (Part 2)
Description: For Part 2, the primary endpoint was to demonstrate that CT-P13 SC is non-inferior to CT-P13 IV, in terms of pharmacokinetics, as determined by the observed Ctrough,week22 (pre-dose level at Week 22).
Time Frame: Week 22
Population: The PK Population consisted of all-randomized population who received at least one full dose of study drug at Week 6 or thereafter, and who had at least one PK result after Week 6 treatment. The primary PK endpoint was analyzed in patients who received all doses (full) of study drug up to Week 22 (prior to Week 22) in the PK population.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: μg/mL
Arm/Group | Arm 1: CT-P13 SC 120/240 mg (Part 2) | Arm 2: CT-P13 IV 5 mg/kg (Part 2)
Number analyzed (Participants) | 59 | 57
μg/mL | 20.9844 [15.2173 to 28.9372] | 1.8181 [1.3054 to 2.5324]
Statistical Analysis 1: Comparison: Arm 1: CT-P13 SC 120/240 mg (Part 2); Primary PK analysis was analyzed using an ANCOVA with treatment as fixed effect and current use of treatment with azathioprine (AZA) or 6-mercaptopurine (6-MP) or methotrexate (MTX) (used or not used), disease (CD or UC), clinical response at Week 6 (responder or non-responder by Clinical Disease Activity Index [CDAI]-70 for CD or partial Mayo score for UC), body weight at Week 6 (<80 kg or ≥80 kg) fitted as covariates; Test type: Non-Inferiority — The non-inferiority of CT-P13 SC to CT-P13 IV was to be concluded if the lower bound of two-sided 90% CI for the ratio of geometric least square means was higher than 80%; Ratio of Geometric LS means = 1154.17, 90% CI 2-sided [786.37 to 1694.00] — The geometric lease square (LS) means, ratio of geometric LS means (CT-P13 SC 120/240 mg to CT-P13 IV 5 mg/kg), and 2-sided 90% CI were obtained from the ANCOVA model

3. Secondary Outcome: Descriptive Statistics for Actual Value of Crohn's Disease Activity Index (CDAI) Score (Part 2 - CD)
Description: For evaluation of efficacy, the secondary endpoint was defined as descriptive statistics for actual value of CDAI score up to Week 54 between the CT-P13 SC and CT-P13 IV treatment groups in active CD patients. The total CDAI scores range from 0 to over 600 with higher scores indicating increased severity of disease. The index is the sum of 8 components multiplied by the relevant weight factor; number of liquid or very soft stools (x2), abdominal pain (x5), general well-being (x7), CD complications (x20), taking lomotil/opiates for diarrhea (x30), abdominal mass (x10), deviation of hematocrit (x6), and percentage deviation from standard weight (x1). Efficacy assessments were done prior to each study drug administrations. Results up to Week 6 in both arms represent efficacy resulting from CT-P13 IV (5 mg/kg) loading dose treatment.
Time Frame: up to Week 54
Population: The efficacy population consisted of the all randomly assigned patients who received at least 1 full dose of study drug (CT-P13 SC or CT-P13 IV) at Week 6 or thereafter and who had at least 1 efficacy evaluation result after Week 6 treatment. All patients in the efficacy population were analyzed according to the treatment they received.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1: CT-P13 SC 120/240 mg (Part 2) | Arm 2: CT-P13 IV 5 mg/kg (Part 2)
Number analyzed (Participants) | 28 | 25
scores on a scale
  Baseline | 296.38 (59.212) | 294.75 (59.899)
  Week 2: number analyzed (Participants) | 28 | 24
  Week 2 | 194.89 (74.943) | 191.03 (79.250)
  Week 6 | 164.99 (96.360) | 144.94 (80.123)
  Week 14: number analyzed (Participants) | 27 | 25
  Week 14 | 136.29 (85.918) | 131.47 (71.444)
  Week 22: number analyzed (Participants) | 24 | 21
  Week 22 | 106.55 (80.461) | 105.08 (60.970)
  Week 30: number analyzed (Participants) | 24 | 20
  Week 30 | 103.81 (88.435) | 106.44 (67.705)
  Week 54: number analyzed (Participants) | 22 | 18
  Week 54 | 92.03 (77.622) | 79.05 (58.960)

4. Secondary Outcome: Proportion of Patients Achieving Clinical Response According to CDAI-100 Criteria (Part 2 - CD)
Description: For evaluation of efficacy, the secondary endpoint was defined as proportion of patients achieving clinical response according to CDAI-100 criteria up to Week 54 between the CT-P13 SC and CT-P13 IV treatment groups in active CD patients. Efficacy assessments were done prior to each study drug administrations. Results up to Week 6 in both arms represent efficacy resulting from CT-P13 IV (5 mg/kg) loading dose treatment.
  Responder according to CDAI-100 criteria was defined as a decrease in CDAI score of 100 points or more from the baseline value.
Time Frame: up to Week 54
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: CT-P13 SC 120/240 mg (Part 2) | Arm 2: CT-P13 IV 5 mg/kg (Part 2)
Number analyzed (Participants) | 28 | 25
Participants
  Week 2 | 13 | 9
  Week 6 | 16 | 17
  Week 14 | 19 | 18
  Week 22 | 21 | 20
  Week 30 | 19 | 16
  Week 54 | 18 | 16

5. Secondary Outcome: Descriptive Statistics for Actual Value of Partial Mayo Score (Part 2 - UC)
Description: For evaluation of efficacy, the secondary endpoint was defined as descriptive statistics for actual value of partial Mayo score up to Week 54 between the CT-P13 SC and CT-P13 IV treatment groups in active UC patients. The partial Mayo scores range from 0-9 with higher scores indicating increased severity of disease. The index is sum of the 3 subscores, each which range from 0 to 3; stool frequency, rectal bleeding and physician's global assessment. Efficacy assessments were done prior to each study drug administrations. Results up to Week 6 in both arms represent efficacy resulting from CT-P13 IV (5 mg/kg) loading dose treatment.
Time Frame: up to Week 54
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1: CT-P13 SC 120/240 mg (Part 2) | Arm 2: CT-P13 IV 5 mg/kg (Part 2)
Number analyzed (Participants) | 38 | 39
scores on a scale
  Baseline | 5.4 (1.31) | 5.9 (1.21)
  Week 2 | 3.3 (2.18) | 3.3 (1.82)
  Week 6 | 2.6 (2.13) | 2.5 (1.74)
  Week 14: number analyzed (Participants) | 36 | 39
  Week 14 | 1.7 (1.62) | 2.3 (1.92)
  Week 22: number analyzed (Participants) | 35 | 36
  Week 22 | 1.3 (1.63) | 2.3 (1.97)
  Week 30: number analyzed (Participants) | 35 | 36
  Week 30 | 1.2 (1.59) | 1.9 (1.88)
  Week 54: number analyzed (Participants) | 32 | 32
  Week 54 | 0.9 (1.31) | 1.0 (1.60)

6. Secondary Outcome: Proportion of Patients Achieving Clinical Response According to the Partial Mayo Score (Part 2 - UC)
Description: For evaluation of efficacy, the secondary endpoint was defined as proportion of patients achieving clinical response according to the partial Mayo score up to Week 54 between the CT-P13 SC and CT-P13 IV treatment groups in active UC patients. Efficacy assessments were done prior to each study drug administrations. Results up to Week 6 in both arms represent efficacy resulting from CT-P13 IV (5 mg/kg) loading dose treatment.
  Responder according to partial Mayo score was defined as a decrease from baseline in partial Mayo score of at least 2 points, with an accompanying decrease in the subscore for rectal bleeding of at least 1 point or an absolute subscore for rectal bleeding of 0 or 1.
Time Frame: up to Week 54
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1: CT-P13 IV 5 mg/kg (Part 2): Each participant received 2 CT-P13 IV infusions with a 2-week interval at Weeks 0 and 2. Then, this group received CT-P13 IV 5 mg/kg (Infliximab) by IV infusion with a 8-week interval from Week 6 up to Week 22 (Weeks 6, 14 and 22). CT-P13 IV was switched to either 120 mg or 240 mg of CT-P13 SC treatment based on their body weight at Week 30 (CT-P13 SC 120 mg for patients < 80 kg; CT-P13 SC 240 mg for patients ≥ 80 kg), and further doses with CT-P13 SC were given up to Week 54.
Arm/Group | Arm 1: CT-P13 SC 120/240 mg (Part 2) | Arm 1: CT-P13 IV 5 mg/kg (Part 2)
Number analyzed (Participants) | 38 | 39
Participants
  Week 2 | 20 | 25
  Week 6 | 28 | 31
  Week 14 | 30 | 33
  Week 22 | 32 | 30
  Week 30 | 33 | 29
  Week 54 | 31 | 28

7. Secondary Outcome: Descriptive Statistics of Observed Ctrough (Trough Concentration [Before the Next Study Drug Administration]) of Infliximab (Part 2)
Description: For evaluation of pharmacokinetics (PK), the secondary endpoint was defined as the analysis of trough concentration of infliximab up to Week 54. The samples were collected at Weeks 0, 2 and 6, and every 8 weeks up to Week 54. During PK monitoring visit (Weeks 22-30), samples were collected every 2 weeks according steady state PK sampling time point. All enrolled patient received CT-P13 IV infusions at Weeks 0 and 2. Patients in SC group were administered with CT-P13 SC at Week 6 and every 2 weeks thereafter up to Week 54. Patients in IV group were administered with CT-P13 IV at Week 6 and every 8 weeks thereafter up to Week 22. Then, CT-P13 IV was switched to CT-P13 SC at Week 30, and further doses with CT-P13 SC were given up to Week 54. No PK results were obtained at Weeks 6 and 14 for SC group and Weeks 12, 20, 24, 26 and 28 for IV group due to 2 weeks and 8 weeks dosing interval, respectively. All patients in PK population were analyzed according to the treatment they received.
Time Frame: up to Week 54
Population: The PK population consisted of the all-randomized population who received at least one full dose of study drug at Week 6 or thereafter and who had at least one PK concentration result after Week 6 treatment.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Arm 1: CT-P13 SC 120/240 mg (Part 2) | Arm 2: CT-P13 IV 5 mg/kg (Part 2)
Number analyzed (Participants) | 63 | 64
μg/mL
  Week 0 | 23.5432 (8.43542) | 21.8589 (7.36954)
  Week 2 | 15.4736 (9.15888) | 14.0747 (7.74070)
  Week 6: number analyzed (Participants) | 0 | 64
  Week 6 |  | 3.7865 (2.99669)
  Week 12: number analyzed (Participants) | 63 | 0
  Week 12 | 20.9700 (9.21851) |
  Week 14: number analyzed (Participants) | 0 | 57
  Week 14 |  | 2.9317 (2.60859)
  Week 20: number analyzed (Participants) | 59 | 0
  Week 20 | 21.4500 (9.86306) |
  Week 22: number analyzed (Participants) | 28 | 48
  Week 22 | 19.6786 (8.94416) | 2.4273 (2.49468)
  Week 24: number analyzed (Participants) | 29 | 0
  Week 24 | 20.1528 (10.53981) |
  Week 26: number analyzed (Participants) | 30 | 0
  Week 26 | 22.3410 (9.81672) |
  Week 28: number analyzed (Participants) | 49 | 0
  Week 28 | 21.0978 (8.98618) |
  Week 36: number analyzed (Participants) | 59 | 53
  Week 36 | 22.1927 (9.97943) | 18.5974 (11.41166)
  Week 44: number analyzed (Participants) | 56 | 50
  Week 44 | 22.5780 (11.72637) | 19.6401 (10.48885)
  Week 52: number analyzed (Participants) | 53 | 49
  Week 52 | 22.7928 (13.17095) | 20.5784 (12.45367)

8. Secondary Outcome: Descriptive Statistics for Actual Value in Fecal Calprotectin Concentration (Pharmacodynamic Parameter) (Part 2)
Description: For evaluation of pharmacodynamic (PD), the secondary endpoint was defined as concentration of Fecal Calprotectin (FC) between 2 treatment groups up to Week 54. The fecal samples for FC were collected at Weeks 0, 2 and 6, and every 8 weeks up to Week 54. All enrolled patients received CT-P13 IV infusions at Weeks 0 and 2. Then, patients in CT-P13 SC group were administered with CT-P13 SC at Week 6 and every 2 weeks thereafter up to Week 54. Patients in the CT-P13 IV group were administered with CT-P13 IV at Week 6 and every 8 weeks thereafter up to Week 22 (Weeks 14 and 22). And then, CT-P13 IV was switched to CT-P13 SC based on body weight at Week 30, and further doses with CT-P13 SC were given up to Week 54. All patients in the PD population were analyzed according to the treatment they received.
Time Frame: up to Week 54
Population: PD population - The PD population consisted of all randomly assigned patients who received at least 1 full dose of study drug (CT-P13 SC, CT-P13 IV) at Week 6 or thereafter, and who had at least 1 PD result after Week 6 treatment.
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | Arm 1: CT-P13 SC 120/240 mg (Part 2) | Arm 2: CT-P13 IV 5 mg/kg (Part 2)
Number analyzed (Participants) | 66 | 64
μg/g
  Baseline | 2094.2 (4114.17) | 2605.2 (8757.77)
  Week 2: number analyzed (Participants) | 62 | 61
  Week 2 | 697.0 (903.85) | 455.0 (561.73)
  Week 6: number analyzed (Participants) | 58 | 62
  Week 6 | 735.3 (1329.11) | 567.3 (956.14)
  Week 14: number analyzed (Participants) | 60 | 62
  Week 14 | 567.6 (751.53) | 706.1 (968.00)
  Week 22: number analyzed (Participants) | 48 | 52
  Week 22 | 796.8 (1950.69) | 1137.0 (2510.62)
  Week 30: number analyzed (Participants) | 49 | 56
  Week 30 | 555.8 (1032.33) | 603.1 (905.60)
  Week 38: number analyzed (Participants) | 56 | 50
  Week 38 | 556.8 (1845.66) | 505.3 (866.04)
  Week 46: number analyzed (Participants) | 56 | 48
  Week 46 | 354.2 (628.37) | 552.2 (1451.62)
  Week 54: number analyzed (Participants) | 49 | 45
  Week 54 | 484.1 (1216.95) | 256.2 (520.12)

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) and treatment emergent serious adverse events (TESAEs) were assessed from the date the informed consent form was signed until the last assessment date or End-of-Study (EOS) visit.
Description: The investigator was responsible for reporting all AEs that were observed or reported during the study, regardless of their relationship to the study drug or clinical significance. Treatment emergent adverse events were pre-specified to only report the most severe event if the same events were occurred to the same patient. All patients who received at least 1 (partial or full) dose of study drug at Week 6 or thereafter were included in safety analysis.
Groups:
- Arm 2: CT-P13 IV 5 mg/kg (Part 2): Each participant received 2 CT-P13 IV infusions with a 2-week interval at Weeks 0 and 2. Then, this group received CT-P13 IV 5 mg/kg (Infliximab) by IV infusion with a 8-week interval from Week 6 up to Week 22 (Weeks 6, 14 and 22). CT-P13 IV were switched to either 120 mg or 240 mg of CT-P13 SC treatment based on their body weight at Week 30, and further doses with CT-P13 SC were given up to Week 54 (CT-P13 SC 120 mg for patients < 80 kg; CT-P13 SC 240 mg for patients ≥ 80 kg).
Arm/Group | Cohort 1: CT-P13 IV 5 mg/kg (Part 1) | Cohort 2: CT-P13 SC 120 mg (Part 1) | Cohort 3: CT-P13 SC 180 mg (Part 1) | Cohort 4: CT-P13 SC 240 mg (Part 1) | Arm 1: CT-P13 SC 120/240 mg (Part 2) | Arm 2: CT-P13 IV 5 mg/kg (Part 2)
All-Cause Mortality (participants affected / at risk) | 1/13 | 0/11 | 1/12 | 0/8 | 0/66 | 0/65
Serious Adverse Events (participants affected / at risk) | 4/13 | 2/11 | 1/12 | 3/8 | 6/66 | 8/65
Other Adverse Events (participants affected / at risk) | 10/13 | 9/11 | 8/12 | 7/8 | 42/66 | 36/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: CT-P13 IV 5 mg/kg (Part 1) (N=13) | Cohort 2: CT-P13 SC 120 mg (Part 1) (N=11) | Cohort 3: CT-P13 SC 180 mg (Part 1) (N=12) | Cohort 4: CT-P13 SC 240 mg (Part 1) (N=8) | Arm 1: CT-P13 SC 120/240 mg (Part 2) (N=66) | Arm 2: CT-P13 IV 5 mg/kg (Part 2) (N=65)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Disseminated tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia legionella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sudden cardiac death (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abscess intestinal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: CT-P13 IV 5 mg/kg (Part 1) (N=13) | Cohort 2: CT-P13 SC 120 mg (Part 1) (N=11) | Cohort 3: CT-P13 SC 180 mg (Part 1) (N=12) | Cohort 4: CT-P13 SC 240 mg (Part 1) (N=8) | Arm 1: CT-P13 SC 120/240 mg (Part 2) (N=66) | Arm 2: CT-P13 IV 5 mg/kg (Part 2) (N=65)
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 4 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 5 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 6 | 2
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4 | 8
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 5 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 6 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 6 | 1
Localized Injection site reaction (General disorders) | 0 | 1 | 3 | 1 | 15 | 3 — General disorders and administration site conditions; preferred term reported as injection site reaction
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 2
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 5 | 4
Headache (Nervous system disorders) | 0 | 0 | 0 | 2 | 5 | 8
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 5 | 5
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 1 | 2 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 2
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bundle branch block right (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 1 | 0 | 3
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Latent tuberculosis (Infections and infestations) | 0 | 0 | 2 | 1 | 1 | 2
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 1
Sinobronchitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0 | 1 | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0
Varicella (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 4 | 2 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 3 — Infusion related reaction occurred between start of administration and 24 hours from the end of IV infusion
Delayed hypersensitivity (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 3 | 0 — Delayed hypersensitivity occurred after 24 hours from the study drug administration
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 0
Blood pressure decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hyperaemia (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 0 | 3 | 1
Pyrexia (General disorders) | 2 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/52/NCT02883452/Prot_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (Part 1) (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT02883452/SAP_001.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (Part 2) (2019-10-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT02883452/SAP_002.pdf